CLINICAL TRIAL: NCT06094088
Title: Examining the Impact of Heated and Non-Heated Yoga on Depression
Brief Title: Researching Heat and Yoga for Mood Enhancement
Acronym: RHYME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Tiny Blue Dot Foundation (Other)
Responsible Party: Principal Investigator, Maren Nyer, Clinical Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023p001916
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heated Yoga (Experimental): The heated (i.e., ~105°F with 40% humidity) yoga will be 90 minutes long and consist of 26 Hatha yoga postures and 2 breathing exercises. The class starts with standing postures for approximately 45-50 minutes, followed by a 2-minute savasana (or corpse pose on the floor) and the remainder of the 90-minute class is completed on the mat. All yoga teachers will be heated yoga certified.
  Interventions: Behavioral: Heated Yoga
- Non-heated Yoga (Active Comparator): The non-heated (i.e., room temperature < 80°F) yoga will be 90 minutes long and consist of 26 Hatha yoga postures and 2 breathing exercises. The class starts with standing postures for approximately 45-50 minutes, followed by a 2-minute savasana (or corpse pose on the floor) and the remainder of the 90-minute class is completed on the mat. All yoga teachers will be heated yoga certified.
  Interventions: Behavioral: Non-Heated Yoga

INTERVENTIONS:
Behavioral: Heated Yoga — Heated yoga described in arm/group description
  Arms: Heated Yoga
Behavioral: Non-Heated Yoga — Non-heated yoga described in arm/group description
  Arms: Non-heated Yoga

SUMMARY:
This study will examine how doing heated yoga or non-heated yoga affects depression.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of heated and non-heated yoga on depressive symptoms. Previous research trials using heated and non-heated yoga interventions have shown promising results for reducing depression and its related outcomes. However, no studies have directly compared the effects of heated vs. non-heated yoga for depression. The researchers aim to address this gap by conducting a non-inferiority trial comparing heated yoga and non-heated yoga interventions to improve depressive symptoms. Both the heated and non-heated yoga interventions will be conducted in-person by certified yoga instructors. Eligible participants will be adults who do not regularly practice yoga or meditation and are experiencing moderate levels of depression. Assessments will be conducted at baseline, mid-treatment, post-treatment, and follow-up using a secure data capture system.

ELIGIBILITY:
Inclusion Criteria:

1. adults (18-65 years old)
2. able to provide consent
3. are able to read and understand English
4. PHQ-9 score between 10-20, indicating moderate but not severe depressive symptom severity (27)
5. Must have filled out the waiver for the community-based yoga studio prior to enrolling in the study.

Exclusion Criteria:

1. have had a bone fracture or joint surgery in the past 6 months
2. not able to walk freely or without difficulty
3. have severe heart failure or lung disease
4. participants endorse an item on the revised Physical Activity Readiness Questionnaire (PAR-Q+) and do not have approval from their treating physician (we will check in with treating physician in the event that participants endorse any item on the PAR-Q+)
5. participants must have a physician responsible for their medical care
6. are pregnant or planning to become pregnant
7. no more than 6 yoga classes in the past 6 months
8. have active suicidal thinking (i.e., PHQ-9 item 9 ≥1 and a positive response to C-SSRS screener items 3, 4, 5, or 6)
9. report manic symptoms (Altman Self-Rating Mania Scale score ≥ 6 (28))
10. are on medications that make dehydration more likely (e.g., lithium, antipsychotics, insulin-dependent)
11. active eating disorders or substance use disorders within the past 12 months
12. antidepressant or psychiatric medications that are initiated less than 8 weeks or a dose change less than 4 weeks prior to screening visit
13. psychotherapy that has been initiated within the past 3 months
14. willingness to keep psychiatric medications and psychotherapy stable throughout the course of the study
15. psychiatric hospitalization within the past year
16. diagnosed with any neurological disorders that would impact participation or make participation unsafe
17. are currently in any active ketamine, ECT, or TMS
18. are unable to follow the study procedures (e.g., not able to travel to the heated or non-heated yoga studios)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Weeks 0, 4, 8, and 20
  This measure is a 9-item self-report questionnaire that is widely used to assess depression symptom severity. PHQ-9 scores range from 0 to 27. A PHQ-9 score ≥10 has a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively.

SECONDARY OUTCOMES:
The World Health Organization-5 Well-Being Index (WHO-5) | Weeks 0, 4, 8, and 20
  This measure is a 5-item self-report questionnaire with positively-worded statements related to positive mood, vitality, and general interest over the prior two weeks. The WHO-5 is reliable, has shown strong construct validity as a measure of general quality of life, and is sensitive to change. The WHO-5 has a score range of 0 to 25, with higher scores indicating better wellbeing.
Patient Reported Outcomes Measurement Information System-29 (PROMIS-29) | Weeks 0, 4, 8, and 20
  This measure has seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, social functioning, sleep disturbance). The scale includes four items per domain, each scored from 1 to 5. The scale also includes one question at the end about pain intensity, which is scored from 0 to 10. The possible score for each domain ranges from 4 to 20 and the total possible score for the entire measure ranges from 28 to150. Higher scores indicate poorer outcomes.
Ruminative Responses Scale (RRS) | Weeks 0, 4, 8, and 20
  This measure is a 22-item questionnaire, commonly used to assess rumination. Items are scored from 1 to 4, the scale has a possible range of 22 to 88, and higher scores indicate poorer outcomes (i.e. higher rumination).
The Five Facet Mindfulness Questionnaire (FFMQ-15) | Weeks 0, 4, 8, and 20
  A self-report instrument that measures mindfulness; derived from factor analytic study of five independent mindfulness questionnaires. The scale contains 39 items, split into five domains (Observing, Describing, Acting with Awareness, Nonjudging, Nonreactivity), with each item being rated from 1 to 5. Some items are reverse coded. Total FFMQ scores range from 39 to 195, with greater scores indicating better outcomes (i.e. greater mindfulness).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orange Door Collaborative, Cambridge, Massachusetts
  - Breathe Yoga Studio, Cambridge, Massachusetts